CLINICAL TRIAL: NCT00003377
Title: A Phase I Study of Extended Field Radiation Therapy With Concomitant Paclitaxel and Cisplatin Chemotherapy in Patients Cervical Carcinoma Metastatic to the Para-Aortic Lymph Nodes
Brief Title: Radiation Therapy, Paclitaxel, and Cisplatin in Treating Patients With Cancer of the Cervix
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Gynecologic Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: GOG Foundation (Network)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000066371; GOG-9804
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Results first posted 2013-02-04 (Estimated); Last update posted 2013-02-04 (Estimated); Status verified 2012-12

CONDITIONS: Cervical Cancer
Keywords: stage III cervical cancer; stage IVA cervical cancer; cervical squamous cell carcinoma; cervical adenocarcinoma; cervical adenosquamous cell carcinoma
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Cisplatin; Paclitaxel; Brachytherapy; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Radiation therapy plus concurrent weekly chemotherapy (Other)
  Interventions: Drug: cisplatin; Drug: paclitaxel; Radiation: brachytherapy; Radiation: radiation therapy

INTERVENTIONS:
Drug: cisplatin
Drug: paclitaxel
Radiation: brachytherapy
Radiation: radiation therapy

SUMMARY:
RATIONALE: Radiation therapy uses high-energy x-rays to damage tumor cells. Paclitaxel and cisplatin may increase the effectiveness of radiation therapy by making the tumor cells more sensitive to the radiation. Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining radiation therapy with chemotherapy may kill more tumor cells.

PURPOSE: This phase I/II trial is studying the side effects and best dose of paclitaxel when given with radiation therapy and cisplatin and to see how well they work in treating patients with cancer of the cervix that has spread to the lymph nodes in the pelvis and abdomen.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the toxicity of extended field radiotherapy with concurrent paclitaxel and cisplatin chemotherapy (as radiation sensitization) in patients with previously untreated carcinoma of the cervix metastatic to the para-aortic lymph nodes.
* Determine the maximum tolerated dose of paclitaxel when combined with cisplatin plus extended field radiotherapy in this patient population.
* Determine the effect of this treatment regimen on progression-free survival, overall survival, and site of recurrence (local vs distant) in these patients.

OUTLINE: This is a multicenter, dose-escalation study of paclitaxel.

Patients receive external beam radiotherapy (RT) to the para-aortic nodes and the pelvis daily for 5 weeks; RT must be completed within 8 weeks of its initiation. During or after external beam RT, intracavitary radiation is administered 1-5 times. Concurrently with external beam RT, patients receive paclitaxel IV over 1 hour followed immediately by cisplatin IV on days 1, 8, 15, 22, 29, and 36.

Cohorts of 3-6 patients receive escalating doses of paclitaxel until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which at least 2 of 6 patients experience dose-limiting toxicity.

Patients are followed every 3 months for 2 years, every 6 months for 3 years, and then annually thereafter or until the time of recurrence or death.

PROJECTED ACCRUAL: A total of 20-40 patients will be accrued for this study within 4 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically proven previously untreated invasive carcinoma of the uterine cervix

  * Squamous cell carcinoma
  * Adenosquamous carcinoma
  * Adenocarcinoma
* TNM classification stage IIIB or IVA (FIGO classification stage IB, IIA, IIB, IIIA, IIIB, or IVA)
* Cytologically or histologically proven metastases to the para-aortic lymph nodes
* No more than 8 weeks since diagnosis
* No metastases to scalene nodes, intraperitoneal metastases, or metastases to other organs outside the radiation field at the time of original clinical and surgical staging

  * Negative CT scan of the chest
* Patients with ureteral obstruction must be treated with stent or nephrostomy tube

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* GOG 0-2

Life expectancy:

* At least 6 months

Hematopoietic:

* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3

Hepatic:

* Bilirubin no greater than 1.5 times normal
* SGOT no greater than 3 times normal

Renal:

* Creatinine less than 2.0 mg/dL
* No renal abnormalities (e.g., pelvic kidney, horseshoe kidney, or renal transplantation) requiring modification of radiation fields

Other:

* Not pregnant
* No septicemia or severe infection
* No other invasive malignancy within the past 3 years except nonmelanoma skin cancer

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* No prior cytotoxic chemotherapy for this or other malignancy

Endocrine therapy:

* Not specified

Radiotherapy:

* No prior radiotherapy for this or other malignancy
* No prior radiotherapy to pelvis or abdomen

Surgery:

* Not specified

Other:

* No other prior therapy for this malignancy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 1999-11; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joan L. Walker, MD, Study Chair — Oklahoma University Cancer Institute
Locations (13):
- United States (13):
  - University of Miami Sylvester Comprehensive Cancer Center, Miami, Florida
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Holden Comprehensive Cancer Center at University of Iowa, Iowa City, Iowa
  - Cancer Institute of New Jersey at the Cooper University Hospital - Voorhees, Camden, New Jersey
  - Comprehensive Cancer Center at Wake Forest University, Winston-Salem, North Carolina
  - MetroHealth's Cancer Care Center at MetroHealth Medical Center, Cleveland, Ohio
  - Cleveland Clinic Cancer Center at Fairview Hospital, Cleveland, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - Arthur G. James Cancer Hospital and Solove Research Institute at Ohio State University, Columbus, Ohio
  - Riverside Methodist Hospital Cancer Care, Columbus, Ohio
  - Oklahoma University Medical Center, Oklahoma City, Oklahoma
  - Cancer Care Associates - Midtown Tulsa, Tulsa, Oklahoma
  - Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania

REFERENCES:
- [Result] Walker JL, Morrison A, DiSilvestro P, von Gruenigen VE; Gynecologic Oncology Group. A phase I/II study of extended field radiation therapy with concomitant paclitaxel and cisplatin chemotherapy in patients with cervical carcinoma metastatic to the para-aortic lymph nodes: a Gynecologic Oncology Group study. Gynecol Oncol. 2009 Jan;112(1):78-84. doi: 10.1016/j.ygyno.2008.09.035. Epub 2008 Nov 17. PMID 19010522

RESULTS

PARTICIPANT FLOW:
Recruitment Details: In Period I 12 patients were treated with weekly cisplatin(30-40 mg/m2) and paclitaxel(30-50 mg/m2) concurrent with extended field radiation. In Period II an additional 17 patients were treated with cisplatin 40 mg/m2 and paclitaxel 40 mg/m2 concurrent with radiation.
Pre-assignment Details: All patients received whole pelvic and extended field radiation at 150 centigray per day for 30 days to the para-aortics, and 180 centigray per day for 25 days to the pelvis.
Groups:
- Arm 1, P I: Cisplatin 40 mg/m2, plus Paclitaxel 30 mg/m2
- Arm 2, P I; Arm 2, P II: Cisplatin 40 mg/m2, plus Paclitaxel 40 mg/m2
- Arm 3, P I: Cisplatin 40 mg/m2, plus Paclitaxel 50 mg/m2
- Arm 4, P I: Cisplatin 30 mg/m2, plus Paclitaxel 50 mg/m2
Period: Period I
Arm/Group | Arm 1, P I | Arm 2, P I | Arm 3, P I | Arm 4, P I | Arm 2, P II
Started | 3 | 3 | 3 | 3 | 0
Completed | 3 | 3 | 2 | 2 | 0
Not Completed | 0 | 0 | 1 | 1 | 0
Not completed — Dose Limiting Toxicity(DLT) | 0 | 0 | 1 | 1 | 0
Period: Period II
Arm/Group | Arm 1, P I | Arm 2, P I | Arm 3, P I | Arm 4, P I | Arm 2, P II
Started | 0 (Patients participated at this dose level only in Period I.) | 0 (Patients participated at this dose level only in Period I.) | 0 (Patients participated at this dose level only in Period I.) | 0 (Patients participated at this dose level only in Period I.) | 17 (All pts enrolled on Per II received cisplatin 40 mg/m2 & paclitaxel 40 mg/m2 concurrent w/ radiation)
Completed | 0 | 0 | 0 | 0 | 16
Not Completed | 0 | 0 | 0 | 0 | 1
Not completed — Ureteral stent complications | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1, P I | Arm 2, P I | Arm 2, P II | Arm 3, P I | Arm 4, P I | Total
Number analyzed (Participants) | 3 | 3 | 17 | 3 | 3 | 29
Age Continuous [Mean (Standard Deviation); unit: years] | 46.4 (13.7) | 54.2 (10.7) | 49.8 (11.0) | 47.6 (8.4) | 47.7 (4.0) | 49.5 (10.1)
Age, Customized [Number; unit: participants]
  20-29 years | 0 | 0 | 1 | 0 | 0 | 1
  30-39 years | 1 | 0 | 1 | 0 | 0 | 2
  40-49 years | 1 | 1 | 9 | 2 | 2 | 15
  50-59 years | 0 | 1 | 2 | 1 | 1 | 5
  60-69 years | 1 | 1 | 4 | 0 | 0 | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 17 | 3 | 3 | 29
  Male | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 3 | 3 | 17 | 3 | 3 | 29
FIGO (International Federation of Gynecology and Obstetrics) Stage [Number; unit: participants] — Clinical staging - Carcinoma of the Cervix Uteri FIGO Classification 1995 specifying invasive carcinoma from Stage 1A (confined to the cervix, identified only microscopically) to Stage 4B (spread to distant organs).
  participants
    1A - disease identified only microscopically | 0 | 0 | 0 | 0 | 0 | 0
    1B - disease confined to cervix | 1 | 1 | 2 | 2 | 0 | 6
    2A - no obvious parametrial involvement | 0 | 0 | 0 | 0 | 0 | 0
    2B - obvious parametrial involvement | 2 | 0 | 4 | 0 | 1 | 7
    3A -disease in lower 3rd of vagina not pelvic wall | 0 | 0 | 0 | 0 | 0 | 0
    3B - disease extended to pelvic wall | 0 | 2 | 7 | 1 | 2 | 12
    4A - disease spread to adjacent organs | 0 | 0 | 4 | 0 | 0 | 4
    4B - disease spread to distant organs | 0 | 0 | 0 | 0 | 0 | 0
Cell Type [Number; unit: participants]
  Adenocarcinoma NOS(not otherwise specified) | 0 | 1 | 1 | 0 | 0 | 2
  Clear cell | 0 | 0 | 0 | 1 | 0 | 1
  Squamous cell | 3 | 2 | 16 | 2 | 3 | 26

OUTCOME MEASURES:

1. Primary Outcome: Dose Limiting Toxicity(DLT)/Significant Dose Delay of Paclitaxel With Cisplatin as Assessed by CTC 2.0 After 6 Cycles of Treatment
Time Frame: up to 21 weeks
Measure: Number; unit: participants
Groups:
- Arm 2, PII: Cisplatin 40 mg/m2, plus Paclitaxel 40 mg/m2
Arm/Group | Arm 1, P I | Arm 2, P I | Arm 3, P I | Arm 4, P I | Arm 2, PII
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 17
participants
  Dose Limiting Toxicity(DLT)/Significant Dose Delay | 0 | 0 | 2 | 2 | 0
  Complications unrelated to treatment | 0 | 0 | 0 | 0 | 1

2. Secondary Outcome: Disease-free Survival at 2 Years
Description: Product-limit estimate of the probability of being alive and progression-free at 24 months based on those 20 patients who were treated at the study recommended dose level (RDL) is 0.65, 95% confidence interval (0.44-0.86).
  Progression is defined as a 50% or greater increase in the product from any lesion documented within eight weeks for study entry or the appearance of any new lesion within eight weeks of entry into study.
Time Frame: 2 years
Measure: Mean (95% Confidence Interval); unit: probability
Groups:
- Arm 2, P I & II: Cisplatin 40 mg/m2, plus Paclitaxel 40 mg/m2
Arm/Group | Arm 2, P I & II
Number analyzed (Participants) | 20
probability | 0.65 [0.44 to 0.86]

3. Secondary Outcome: Overall Survival at 2 Years
Description: Product-limit estimate of the probability of being alive at 24 months based on those 20 patients who were treated at the study recommended dose-level is 0.80, 95 % confidence interval (0.62-0.97)
Time Frame: 2 years
Measure: Mean (95% Confidence Interval); unit: probability
Arm/Group | Arm 2, P I & II
Number analyzed (Participants) | 20
probability | 0.80 [0.62 to 0.97]

ADVERSE EVENTS:
Arm/Group | Arm 1, P I | Arm 2, P I | Arm 3, P I | Arm 4, P I | Arm 2, P II
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3 | 1/3 | 2/3 | 1/17
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 3/3 | 2/3 | 15/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1, P I (N=3) | Arm 2, P I (N=3) | Arm 3, P I (N=3) | Arm 4, P I (N=3) | Arm 2, P II (N=17)
Pulmonary disorders (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea and vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypomagnesia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypocalcemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1, P I (N=3) | Arm 2, P I (N=3) | Arm 3, P I (N=3) | Arm 4, P I (N=3) | Arm 2, P II (N=17)
Neutropenia (Blood and lymphatic system disorders) | 2 | 0 | 1 | 1 | 7
Leukopenia (Blood and lymphatic system disorders) | 2 | 3 | 1 | 1 | 10
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 2
Anemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 1
Pulmonary Embolism (Cardiac disorders) | 0 | 0 | 0 | 1 | 1
Hypotension (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 3
Nausea and vomiting (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 4
Diarrhea (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 3
Vaginal Bleeding (General disorders) | 0 | 0 | 0 | 0 | 1 — CTCAE 2.0 categorized as "Hemorrhage"
Febrile neutropenia (Infections and infestations) | 1 | 0 | 0 | 0 | 3
Hypomagnesia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0 | 0
Hypokalemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 1 | 3
Hypocalcemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 1
Seizure (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Confusion (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Pelvic pain (General disorders) | 0 | 0 | 0 | 0 | 1 — CTCAE 2.0 categorized as "Pain"
Abdominal pain (General disorders) | 0 | 0 | 0 | 0 | 1 — CTCAE 2.0 categorized as "Pain"
ALT (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1
Prothrombin time (Vascular disorders) | 0 | 0 | 0 | 0 | 1 — CTCAE 2.0 categorized as "Coagulation"

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No